CLINICAL TRIAL: NCT06008613
Title: 3D Holographic Guidance, Navigation, and Control (3D GN&C) for Endovascular Aortic Repair (EVAR)
Brief Title: 3D Holographic Guidance, Navigation, and Control for Endovascular Aortic Repair
Acronym: 3D-GN&C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-753; 5R44HL139290-03 (NIH)
Record Dates: First submitted 2023-08-09; First posted 2023-08-23 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: AAA; EVAR
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention (Experimental): Electromagnetic guidance and tracking as an adjunct to and confirmed by fluoroscopic imaging to be used with Cook Zenith Flex AAA Endovascular Graft.
  Interventions: Device: 3D Holographic Guidance, Navigation, and Control (3D GN&C)

INTERVENTIONS:
Device: 3D Holographic Guidance, Navigation, and Control (3D GN&C) — Using electromagnetic (EM) guidance and tracking to precisely place a Cook Zenith Flex AAA bifurcated stent graft during EVAR. EM guidance and tracking is enabled using a system consisting of:
  1. experimental 3D guidance, navigation, and control (3D-GNC) software developed by Centerline Biomedical, Inc., integrated with the company's FDA-cleared Intra-Operative Positioning System (IOPS),
  2. FDA-cleared compatible sensorized guidewires added to the Cook Zenith Flex delivery system, and
  3. 3D visualization on the IOPS mobile cart monitor and 3D holographic visualization overlaid on the patient during the procedure using a head mounted display (HMD), the Microsoft HoloLens 2.

SUMMARY:
This is an Early Feasibility Study to evaluate the usability, safety and functionality of 3D holographic guidance, navigation, and control (3D-GNC) as an adjunct to and confirmed by fluoroscopic imaging to be used with Cook Zenith Flex AAA Endovascular Graft.

DETAILED DESCRIPTION:
The goal of this clinical study is to evaluate the feasibility of using electromagnetic (EM) guidance and tracking to precisely place a Cook Zenith Flex AAA bifurcated stent graft during EVAR. EM guidance and tracking is enabled using a system consisting of the following: 1) experimental 3D guidance, navigation, and control (3D-GNC) software developed by Centerline Biomedical, Inc., integrated with the company's FDA-cleared Intra-Operative Positioning System (IOPS), 2) FDA-cleared compatible sensorized guidewires added to the Cook Zenith Flex delivery system and 3) 3D visualization on the IOPS mobile cart monitor and 3D holographic visualization overlaid on the patient during the procedure using a head mounted display (HMD), the Microsoft HoloLens 2. Planning and execution of each case will be major steps in demonstrating feasibility of the technology beyond non-clinical and preclinical testing.

ELIGIBILITY:
Inclusion Criteria:

1. The patient meets the instructions for use (IFU) for the 24-28 mm body Cook Zenith Flex AAA bifurcated stent graft.

   1. Adequate iliac/femoral access compatible with the required introduction system
   2. Non aneurysmal infrarenal aortic segment (neck) proximal to the aneurysm:

   i. With a length of at least 15mm ii. With a diameter measured outer wall to outer wall of no greater than 26mm and no less than 20mm iii. With an angle less than 60 degrees relative to the long access of the aneurysm and iv. With an angle less than 45 degrees relative to the axis of the suprarenal aorta c. Iliac artery distal fixation site greater than 10mm in length and 7.5-20mm in diameter (measured outerwall to outerwall).
2. Male/female, aged ≥ 18
3. Patient fulfilling criteria for needing endovascular repair of abdominal aortic aneurysm according to routine clinical practice criteria of the participating center
4. Women of childbearing potential must be non-pregnant, non-lactating, and not planning to become pregnant during the course of the trial; and have a negative urine or serum pregnancy test within 7 days prior to index procedure
5. Provide written informed consent as applicable and defined by site country regulation
6. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Contraindications for Cook Zenith Flex Aortic endograft:

   1. Patients with known sensitivities or allergies to stainless steel, polyester, solder (tin, silver), polypropylene, or gold
   2. Patients with a systemic infection who may be at increased risk of endovascular graft infection
2. Presence of electronic implants, e.g., cardiac pacemaker, AICD or nerve stimulator
3. Presence of metallic implants above the knee, e.g., artificial hip
4. Patients not willing or able to give informed consent
5. Pregnant women
6. Patients' inability to have a contrasted CT scan
7. Current or planned participation in any other investigational drug or medical device clinical study that has not completed primary endpoint(s) evaluation;
8. Other medical, social, or psychological issues that in the opinion of the investigator preclude the subjects from receiving this treatment, and the procedures and evaluations pre- and posttreatment
9. Anatomy outside of the IFU for a 24-28 mm Cook Zenith Flex AAA bifurcated stent graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful implantation of Cook Zenith AAA Endovascular Graft using the 3D-GN&C device | During the procedure
  Correct positioning of the endovascular stent graft confirmed by fluoroscopic imaging

SECONDARY OUTCOMES:
Delivery system placement in the intended location | During the procedure
  Distance between the fluoroscopy and digital subtraction angiography (mm)

OTHER OUTCOMES:
Incidence of AE/SAE related to 3D-GN&C device | Through study completion, an average of 30 days
  Incidence of SAE (serious adverse events) related to 3D-GNC device as well as incidence of non-SAE (non-Serious Adverse Events) related to 3D-GNC device

CONTACTS AND LOCATIONS:
Overall Officials: Francis Caputo, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No